CLINICAL TRIAL: NCT00928616
Title: Differential Effects of "Functional Foods" Supplemented With Plant Sterol Esters on Blood Cells and Serum Parameters.
Brief Title: Differential Effects of a Diet Supplementation With Plant Sterol Esters on Human Monocytes
Acronym: PSE-MO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Oliver Weingärtner MD, University of the Saarland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 108/07; 108/07
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Hyperlipidemia
Keywords: hyperlipidemia; plant sterols; monocytes
MeSH Terms: conditions — Hyperlipidemias | interventions — Margarine; Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- plant sterol esters (Experimental): Participants consume plant sterol ester supplemented margarine (3 g/day)
  Interventions: Dietary Supplement: margarine + plant sterol esters
- Placebo (Placebo Comparator): Placebo is a non-sterol ester supplemented margarine
  Interventions: Dietary Supplement: margarine (placebo)

INTERVENTIONS:
Dietary Supplement: margarine + plant sterol esters — margarine supplemented with plant sterol esters (3g/day) over the time period of 4 weeks
  Other Names: plant sterols
  Arms: plant sterol esters
Dietary Supplement: margarine (placebo) — non-sterol ester supplemented margarine
  Other Names: regular margarine
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of a diet supplementation with plant sterol esters on serum lipids, plant sterol concentrations and monocyte subpopulations.

DETAILED DESCRIPTION:
This study investigates effects of a diet supplementation with plant sterol esters on serum lipids, plant sterol concentrations and monocyte subpopulations.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals without known cardiovascular diseases

Exclusion Criteria:

* drugs that interfere with cholesterol metabolism
* other use of dietary supplements
* vegetarianism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
monocyte subpopulations | 4 weeks

SECONDARY OUTCOMES:
serum parameters (lipids, plant sterol concentrations, inflammation parameters) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Weingärtner, MD, Principal Investigator — Universitätsklinikum des Saarlandes, Klinik für Innere Medizin III
Locations (1):
- Universitätsklinikum des Saarlandes, Klinik für Innere Medizin III, Homburg, Saarland, Germany